CLINICAL TRIAL: NCT06622538
Title: Orotracheal Intubation with the ORION Videolaryngoscope Versus the King Vision Videolaryngoscope in Adult Patients Without Predictors of a Difficult Airway
Brief Title: Orotracheal Intubation with the ORION Videolaryngoscope Versus the King Vision Videolaryngoscope in Adult Patients: ORION Trial
Acronym: ORION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Juan Fernando Bautista Garcia, M.D., Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DI/24/310/03/26
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Orotracheal Intubation; Videolaryngoscopes (VL); 3D Printing; Anesthesia
Keywords: 3d printing; Orotracheal intubation; videolaryngoscope; ORION; Additive Manufacturing

STUDY DESIGN:
Intervention Model Description: Randomization in two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videolaryngoscope King Vision (Active Comparator): The King Vision video laryngoscope used in this study has a 45° angulation, with a disposable No. 3 blade and no channel for the orotracheal tube.
  Interventions: Device: Orotracheal intubation
- Videolaryngoscope ORION (Experimental): The ORION video laryngoscope is designed by additive manufacturing, has the same dimensions as a Macintosh No. 3 blade, with 45° angulation, is biocompatible and reusable when subjected to high-level disinfection with 2% Glutaraldehyde for 40 minutes. It has an endoscopic camera fully covered in the body of the videolaryngoscope of 8 mm diameter with 2 megapixels with a resolution of 1280x720, has a viewing angle of 70°, has 6 LEDS with adjustable intensity and the camera has an anti-fogging system and can be connected to any mobile device with Android operating system through a free application. (AN98 Version 2.2.0). It complies with ISO 7376:2020 standards for orotracheal intubation laryngoscopes because its blade withstands a stiffness of more than 60 Newtons and a resistance of more than 150 Newtons.
  Interventions: Device: Orotracheal intubation

INTERVENTIONS:
Device: Orotracheal intubation — Patients who meet the inclusion criteria and sign the informed consent form will be intubated with the ORION or King Vision video laryngoscope according to randomisation.

SUMMARY:
This study aims to compare the ORION video laryngoscope with the King Vision video laryngoscope for orotracheal intubation in patients without predictors of difficult airway scheduled for elective surgery under general anesthesia.

DETAILED DESCRIPTION:
The video laryngoscope, compared to direct laryngoscopy, provides better visualization of the laryngeal and glottic structures, a higher success rate for intubation on the first attempt, and a lower incidence of complications such as mucosal injury, dental injury, and esophageal intubations. Despite the advantages offered by video laryngoscopy, its use is not widespread in developing countries due to high costs. For this reason, the ORION video laryngoscope was developed as a low-cost, reusable device that can undergo high-level disinfection. It is designed using additive manufacturing and meets the standards for biocompatibility, rigidity, and resistance. Additionally, it has undergone preclinical testing in simulation models where anesthesiologists have approved its use in real clinical scenarios. In this study, patients scheduled for elective surgery under general anesthesia without predictors of difficult airway will be included and randomized to be intubated with either the ORION video laryngoscope or the King Vision video laryngoscope. The study will compare the success of intubation on the first attempt, the time taken for intubation, the level of visualization of the glottic structures, and the associated complications between the two video laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age scheduled for elective surgery requiring general anesthesia.
* Patients without predictors of difficult airway.
* Patients with ASA I-II classification.
* Patients with BMI less than 35 kg/mts2.

Exclusion Criteria:

* Pregnant women.
* Patients requiring emergency surgery.
* Patients with chronic obstructive pulmonary disease.
* Patients with a history of chronic ischemic heart disease.
* Patients with a history of asthma.
* Patients who have not signed the informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Successful first attempt | After the endotracheal intubation completed
  Measurement of orotracheal intubations obtained in the first attempt of videolaryngoscopy with the two videolaryngoscopes, successful orotracheal intubation will be corroborated by capnography. Measured in percentage (%).

SECONDARY OUTCOMES:
Intubation time | After the endotracheal intubation completed
  Time elapsed from the time the video laryngoscope blade crosses the dental arch until the orotracheal tube is inserted into the trachea, this time will be measured for each video laryngoscope. Measured in seconds (s).
Laryngeal visualisation measured with the Cormack Lehane scale | After the endotracheal intubation completed
  Measurement of visualization of glottic structures using the Cormack Lehane scale in grade I, II, II and IV obtained with both video laryngoscopes. Measured in percentage (%).
Laryngeal visualisation measured with the POGO scale | After the endotracheal intubation completed
  Measurement of the visualization of the glottic structures using the POGO (Percentage of Glottic Opening) scale from 0% to 100% obtained with both video laryngoscopes. Measured in percentage (%).
Esophageal intubation | After the endotracheal intubation completed
  Measurement of the number of esophageal intubations obtained with both video laryngoscopes. Measured in percentage (%)
Complications | After the endotracheal intubation completed
  Measurement of complications (mucosal, lip, oral, pharyngeal and laryngeal injury, total or partial fracture of a tooth and Hypoxemia) that occur with the use of the ORION and King Vision Videolaryngoscopes. Measured in percent (%)
Number of video laryngoscopy attempts | After the endotracheal intubation completed
  Measurement of the number of video laryngoscopy attempts to successful intubation with both video laryngoscopes. Measurement in percentage (%)
Intubation failure | After the endotracheal intubation completed
  Three videolaryngoscopies with duration of 120 seconds each without achieving orotracheal intubation. The number of intubation failures of both videolaryngoscopes will be measured in percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Fernando Bautista Garcia, Principal Investigator — Hospital General de Mèxico Dr. Eduardo Liceaga
Locations (1):
- Hospital General de Mèxico Dr. Eduardo Liceaga, Mexico City, Cuauhtemoc, Mexico

IPD SHARING:
Plan to Share IPD: No